CLINICAL TRIAL: NCT01551771
Title: A Single-centre, Masked, Placebo-controlled Four Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Repeat Doses of the CC-chemokine Receptor 3 (CCR3) Antagonist, GW824575, Coadministered With or Without Food in Healthy Male Subjects
Brief Title: GW824575 First Time in Human
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 115802
Record Dates: First submitted 2012-02-09; First posted 2012-03-13 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Retinal Diseases
Keywords: CCR3 antagonist
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GW824575 (Experimental): Investigational treatment - Swedish Orange Coloured, opaque hard gelatin capsule
  Interventions: Drug: GW824575 matched-placebo
- GW824575 matched-placebo (Placebo Comparator): Placebo
  Interventions: Drug: GW824575

INTERVENTIONS:
Drug: GW824575 — Investigational treatment - Swedish Orange Coloured, opaque hard gelatin capsule
  Arms: GW824575 matched-placebo
Drug: GW824575 matched-placebo — Placebo
  Arms: GW824575

SUMMARY:
This study is the first administration of GW824575 in humans. This will be a single centre, masked, placebo-controlled study, to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of GW824575, given as single and repeated oral doses to healthy male subjects. The study will be comprised of 4 parts and enroll approximately 40 subjects: Part A will consist of two cohorts of 8 healthy male subjects to assess the safety, tolerability, PK, and PD of ascending single oral doses of GW824575. All available safety, tolerability, and PK data will be monitored prior to each dose escalation. In order to support the possible indication for age-related macular degeneration (AMD), Part B will be one cohort of 12 subjects to examine the safety, tolerability, PK, and PD of a repeated dose of GW824575 over 21 days in healthy male subjects who are greater than or equal to 50 years of age. The total daily dose in this cohort will not exceed the maximum tolerated dose (MTD) from Parts A and D. Subjects in this cohort will undergo ophthalmology assessments before receiving investigational product and after Day 7 of the 21-day in-patient treatment, after steady state has been reached. As part of protocol amendment 2, Part C (Cohort 4) is removed from the protocol. Part D, added under protocol amendment 2, will consist of one cohort of 12 healthy male subjects to assess safety, tolerability, PK, and PD of ascending single doses of GW824575 as well as the effect of food on the PK of GW824575.

DETAILED DESCRIPTION:
Part A will consist of two cohorts of healthy male subjects to assess the safety, tolerability, and PK of ascending single oral doses of GW824575. The sponsor will review available safety, tolerability, and PK data and, where available, PD receptor occupancy (from the eosinophil shape change data) data before each dose escalation. Outcome measures in Part A will be assessed and presented through 48 hours post-dose for each of up to 4 single dose escalations per cohort. Part B will be one cohort to examine the safety, tolerability and PK of a repeated dose of GW824575 over 21 days in healthy male subjects who are greater than or equal to 50 years of age. Subjects in this cohort will undergo ophthalmic assessments before receiving investigational product and after Day 7 of the 21-day in-patient treatment, after steady state has been reached. The PD endpoints such as receptor occupancy will be assessed. The dosing regimen (once or twice daily) will be determined by PK data from Part A; however, regardless of dosing regimen, subjects will only receive a single dose in the morning on Days 1 and 21 of the treatment period. Outcome measures in Part B (Cohort 3) will be assessed and presented through 21 days repeat dosing until 48 hours post-dose last dose (i.e., on Day 23). If a safety signal is noted during, or after, the conduct of Cohort 3 of the study; the cohort may be halted or dose down-titrated, and an additional cohort, at a lower dose, may be instituted in Part B as Cohort 5. Dose selection for the additional cohort (Cohort 5) will be informed by the aggregate safety, PK, and PD data available at that time. Part D will consist of one cohort of healthy male subjects. The cohort will 1) explore the effect of a high fat meal on the PK of GW824575 during two treatment periods with approximately 48 hour washout between periods and 2) assess the safety, tolerability, and PK of ascending single oral doses of GW824575 administered in the fasting state or with a standard meal in up to 3 additional treatment periods with at least 6-day washout between periods. The sponsor will review available safety, tolerability, and PK data and, where available, PD RO (from the eosinophil shape change data) data before each dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* For subjects in Parts A or D - Male subjects between 18 and 65 years of age inclusive, at the time of signing the informed consent.

For subjects in Part B - Male subjects greater than or equal to 50 years of age, at the time of signing the informed consent..

* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in protocol. This criterion must be followed from the time of the first dose of study medication until 4 months post-last dose.
* Body weight greater than or equal to 55 kg and BMI within the range 18 - 31 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTc < 450 msec.
* Normotensive, after having rested quietly in a supine position for at least 15 minutes, with a systolic blood pressure less than or equal to 120 mmHg and diastolic blood pressure less than or equal to 80mmHg and a heart rate less than or equal to 100 beats per minute. Subjects with "pre-hypertension" (systolic blood pressure 121-140 mmHg and diastolic blood pressure 81 to 99mmHg) must be cleared by the medical monitor.
* Willingness and ability to swallow multiple size 00 capsules as part of study participation.
* For subjects in Part B only - Best-corrected visual acuity better than 20/80 (Snellen equivalent; 54 or more ETDRS letters) in both eyes.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Significant infection within 4 weeks prior to the first dosing day.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months (12 weeks), 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and throughout the study, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Any prior intraocular surgery, excluding cataract surgery.
* Any prior eye surgery within three months to first dose of study medication.
* Subjects with glaucoma (controlled or uncontrolled).
* Inability to withhold contact lens wear from the time of the screening ophthalmic assessments until the treatment ophthalmic assessments have been performed (the wearing of glasses is permitted).
* Within 6 months prior to the Screening Visit, use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoxamine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, and ethambutol).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-04-12 (Actual); Study Completion 2012-04-12 (Actual)

PRIMARY OUTCOMES:
Subject tolerability as measured by the number (and frequency) of subjects who experience adverse events after single ascending doses of GW824575 | Parts A and D - Through the expected 48-hour duration of hospital stay.Through the expected 48-hour duration of hospital stay.
  To assess the safety and tolerability of single doses of GW824575 in healthy male subjects.
Subject tolerability as measured by the number (and frequency) of subjects who experience adverse events after repeat doses of GW824575 | Part B through the expected 23-day duration of hospital stay.
  To assess the safety and tolerability of repeat doses of GW824575 in healthy male subjects who are greater than or equal to 50 years of age

SECONDARY OUTCOMES:
Pharmacokinetic parameters such as Cmax, AUC, half-life, Tmax of GW824575 after single dosing. | Parts A and D - predose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours of each hospital stay.
  To characterise the PK profile of single doses of GW824575 in healthy male subjects
Pharmacokinetic parameters such as Cmax, AUC, half-life, Tmax of GW824575 after repeat dosing. | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24, hours on Day 1 of dosing and on Day 21 of dosing in Part B.
  To characterise the PK profile of repeat doses of GW824575 in healthy male subjects who are greater than or equal to 50 years of age
Single dose - eosinophil shape change assay | 24 to 27 hours post dose.
  To determine the PD effect of single doses of GW824575 in healthy male subjects.
Repeat dose - eosinophil shape change assay | Part B at 3, 8 and 24 hours post last dose on Day 21.
  To determine the PD effect of repeat doses of GW824575 in healthy male subjects who are greater than 50 years of age
Urine, serum and bile sampling for GW824575 | Part B (only) at 12-hours after 12 days of repeat dosing.
  To investigate the metabolism of GW824575 following single and repeat doses in healthy male subjects who are greater than or equal to 50 years of age.
Changes in safety laboratory values after single ascending doses of GW824575 | Parts A and D - At the conclusion of the expected 48-hour duration of hospital stay.
  To assess the safety of single dose of GW824575 in healthy male subjects
Changes in safety laboratory values after repeat dosing with GW824575 | Part B through the expected 22-day duration of hospital stay.
  To assess the safety of repeat doses of GW824575 in healthy male subjects who are greater than or equal to 50 years of age

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115802 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115802?search=study&search_terms=115802#rs
- Available data/document: Clinical Study Report: 115802 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115802 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115802 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115802 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115802 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115802 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115802 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register